CLINICAL TRIAL: NCT02489123
Title: Androgen Receptor Targeting in Mantle Cell Lymphoma: A Pilot Trial of Enzalutamide
Brief Title: Enzalutamide in Treating Patients With Relapsed or Refractory Mantle Cell Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Accrual goal not met
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Comprehensive Cancer Network (Network)
Responsible Party: Principal Investigator, Ajay Gopal, Professor, Department of Medicine, Division of Oncology; Director, Hematologic Malignancies Medical Oncology, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9340; NCI-2015-00947 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9340 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH); RG1715046 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2015-06-30; First posted 2015-07-02 (Estimated); Results first posted 2021-08-10 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-07

CONDITIONS: Ann Arbor Stage I Mantle Cell Lymphoma; Ann Arbor Stage II Mantle Cell Lymphoma; Ann Arbor Stage III Mantle Cell Lymphoma; Ann Arbor Stage IV Mantle Cell Lymphoma; Recurrent Mantle Cell Lymphoma; Refractory Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (enzalutamide) (Experimental): Patients receive enzalutamide PO QD. Courses 1-3 repeat every 4 weeks (28 days) and subsequent courses repeat every 12 weeks (84 days) in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Enzalutamide; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Enzalutamide — Given PO
  Other Names: ASP9785; MDV3100; Xtandi
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This pilot clinical trial studies enzalutamide in treating patients with mantle cell lymphoma that has returned after a period of improvement (relapsed) or has not responded to previous treatment (refractory). Androgens can cause the growth of cancer cells. Antihormone therapy, such as enzalutamide, may lessen the amount of androgen made by the body.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Perform a preliminary assessment of the efficacy of single-agent enzalutamide, based on overall response rate, in subjects with relapsed/refractory mantle cell lymphoma (MCL) or previously untreated MCL.

SECONDARY OBJECTIVES:

I. To evaluate the duration of disease control (progression free survival) in patients with MCL treated with enzalutamide.

II. To evaluate the safety profile of enzalutamide in MCL.

III. To gain preliminary data on clinical activity and toxicity of this regimen in male versus (vs.) female patients.

OUTLINE:

Patients receive enzalutamide orally (PO) once daily (QD). Courses 1-3 repeat every 4 weeks (28 days) and subsequent courses repeat every 12 weeks (84 days) in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed relapsed/refractory or previously untreated mantle cell lymphoma (any stage)
* Patients with untreated MCL should be asymptomatic or minimally symptomatic from their MCL and without aggressive clinicopathological features that would otherwise warrant immediate intensive therapy; these will generally be patients who qualify for an initial period of "watch and wait" per clinical discretion
* Patients must have metabolically active (positron emission tomography [PET] scan positive) measurable disease (defined as lesions greater than 1.5 cm long axis that can be accurately measured in two dimensions by computed tomography [CT])
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Absolute neutrophil count (ANC) >= 1000/mm^3 or >= 750/mm^3 in the setting of marrow involvement by disease (independent of growth factor or transfusion support)
* Platelets >= 50,000/mm^3 or >= 30,000/mm^3 in the setting of marrow involvement by disease or splenomegaly due to disease (independent of growth factor or transfusion support)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3 x upper limit of normal (ULN)
* Total bilirubin =< 1.5 x ULN unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin
* Creatinine clearance (CrCl) >= 30 mL/min (as calculated by Cockcroft-Gault equation)
* All patients must be informed of the investigational nature of this study and have given written consent in accordance with institutional and federal guidelines; patient must sign an informed consent document indicating that they understand the purpose of and procedures required for the study, and are willing to participate in and comply with the guidelines of the study
* Women of childbearing potential and men who are sexually active must affirm they are practicing a highly effective method of barrier birth control during and after the study consistent with local regulations regarding the use of birth control methods for subjects participating in clinical trials; men must agree to not donate sperm during or after the study; these restrictions apply throughout the treatment period and for three months after the last dose of enzalutamide
* Women of childbearing potential must have a negative serum (beta-human chorionic gonadotropin [beta-hCG]) or urine pregnancy test at screening; women who are pregnant or breastfeeding are ineligible for this study

Exclusion Criteria:

* Uncontrolled illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements within 6 months of enrollment
* Known active central nervous system lymphoma
* Known clinically significant heart disease as evidenced by:

  * Myocardial infarction within 6 months of enrollment
  * Uncontrolled angina within 6 months of enrollment
  * Congestive heart failure New York Heart Association (NYHA) class III or IV, or a history of congestive heart failure NYHA class III or IV in the past, unless a screening echocardiogram (ECHO) or multi-gated acquisition scan (MUGA) within 3 months results in a left ventricular ejection fraction >= 45%
  * Clinically significant ventricular arrhythmias
  * History of Mobitz II second degree or third degree heart block without a permanent pacemaker in place
  * Bradycardia as indicated by a heart rate < 50 beats per minute at screening visit
  * Hypotension as indicated by systolic blood pressure (SBP) =< 85 on 2 consecutive measurements at screening visit
  * Uncontrolled hypertension as indicated by SBP > 170 mmHg or diastolic blood pressure (DBP) > 105 mmHg on 2 consecutive measurements at screening visit
* Child Pugh class C hepatic dysfunction
* History of seizures
* Any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of enzalutamide, or put the study outcomes at undue risk
* Patients with other prior malignancies except for adequately treated basal cell carcinoma, squamous cell carcinoma of the skin, breast or cervical cancer in situ, or other cancer from which the patient has been disease-free for 5 years or greater, unless approved by the protocol investigator / lead-sub-investigator
* Chemotherapy, immunotherapy, biologically targeted therapy, other investigational agent, or radiation therapy within 3 weeks of initiation of enzalutamide therapy; for patients with objectively progressive disease on a Bruton tyrosine kinase (BTK)-targeting agent whom in the opinion of the investigator would not tolerate a 21 day washout period, a > 5 half-lives washout period will be allowed
* Prior allogeneic transplant with graft-versus-host disease (GVHD) requiring ongoing immunosuppressive therapy
* Human immunodeficiency virus (HIV)-positive individuals on combination antiretroviral therapy are ineligible
* Ongoing treatment with hormonal agents (e.g. finasteride, dutasteride, ketoconazole, hormonal birth control, estrogen replacement therapy, testosterone replacement therapy) or herbal products that may have hormonal activity (saw palmetto, black cohosh); patients taking these agents are eligible for screening, but must be willing to undergo a washout period of 4 weeks prior to starting study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-08-11 (Actual); Primary Completion 2020-06-16 (Actual); Study Completion 2020-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Gopal, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Enzalutamide)
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Enzalutamide)
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 2
Age, Continuous [Median (Full Range); unit: Years] | 60 [47 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response Rate (ORR) Including Complete Response (CR) and Partial Response (PR) as Measured by Standard Criteria
Description: An ORR of 20% (4 or more responses among 20 patients) will be taken as a benchmark for success for the primary endpoint of this pilot study. Evaluation of response is per standard NCI Response Criteria Cheson 2014 and assessed by PET-CT; CR = complete metabolic response, PR = decrease by more the 50% in the sum of the product of the perpendicular diameters.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Enzalutamide)
Number analyzed (Participants) | 7
Participants | 0

2. Secondary Outcome: Time to Treatment Failure
Time Frame: From the first treatment administration to the first time to treatment failure, assessed up to 5 years
Measure: Median (Full Range); unit: Weeks
Arm/Group | Treatment (Enzalutamide)
Number analyzed (Participants) | 8
Weeks | 14 [10 to 35]

3. Secondary Outcome: Progression-free Survival
Description: Kaplan-Meier methodology will be used to estimate event-free curves and corresponding quartiles (including the median).
Time Frame: From first study drug administration to the first occurrence of disease progression or death from any cause, assessed up to 5 years
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment (Enzalutamide)
Number analyzed (Participants) | 8
Months | 4.1 [1.3 to 8.3]

4. Secondary Outcome: Overall Survival
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Enzalutamide)
Number analyzed (Participants) | 8
Participants | 4

5. Secondary Outcome: Number of Participants With One or More Adverse Events, Measured by National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0
Time Frame: Up to 30 days after study treatment completion, an average of 18 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Enzalutamide)
Number analyzed (Participants) | 8
Participants | 8

6. Secondary Outcome: Disease Control Rate (CR + PR + Stable Disease [SD] > 3 Months)
Description: The count of participants who achieved a CR, PR, or SD for greater than 3 months.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Enzalutamide)
Number analyzed (Participants) | 8
Participants | 4

ADVERSE EVENTS:
Time Frame: Adverse Events of Grade 3 and above will be monitored and recorded from the time of the first dose of study treatment through 30 days following the end of study treatment, an average of 18 weeks.
Arm/Group | Treatment (Enzalutamide)
All-Cause Mortality (participants affected / at risk) | 4/8
Serious Adverse Events (participants affected / at risk) | 1/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Enzalutamide) (N=8)
Triple Arthrodesis Right Ankle Surgery (Musculoskeletal and connective tissue disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Enzalutamide) (N=8)
Abdominal Pain (Gastrointestinal disorders) | 2 (2)
Agitation (Psychiatric disorders) | 2 (3)
Decreased Urination (Renal and urinary disorders) | 2 (2)
Breast Tenderness (Reproductive system and breast disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hot Flashes (Vascular disorders) | 5 (6)
Platelet Count Decreased (Investigations) | 1 (1)
Fatigue (General disorders) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)
Headache (Nervous system disorders) | 1 (1)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Constipation (Gastrointestinal disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1)
Ankle Pain (General disorders) | 1 (3)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Decrease in genital size (Reproductive system and breast disorders) | 1 (1)
Genital oder (General disorders) | 1 (1)
Skin Changes (Skin and subcutaneous tissue disorders) | 3 (3)
Non-cardiac chest pain (General disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 1 (1)
Eye Pain (Eye disorders) | 1 (1)
Increased white blood cell count (Blood and lymphatic system disorders) | 1 (1)
Paresthesia (Skin and subcutaneous tissue disorders) | 1 (1)
Nail Ridging (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-26): https://cdn.clinicaltrials.gov/large-docs/23/NCT02489123/Prot_SAP_000.pdf